CLINICAL TRIAL: NCT00457808
Title: Rapamycin Therapy of Angiomyolipomas in Patients With Tuberous Sclerosis Complex and Sporadic Lymphangioleiomyomatosis
Brief Title: Rapamycin Therapy for Patients With Tuberous Sclerosis Complex and Sporadic LAM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: The LAM Foundation (Other); Tuberous Sclerosis Alliance (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCHMC IRB # 02-10-16; R21CA103486 (NIH)
Record Dates: First submitted 2007-04-06; First posted 2007-04-09 (Estimated); Last update posted 2007-04-09 (Estimated); Status verified 2007-04

CONDITIONS: Tuberous Sclerosis; Lymphangioleiomyomatosis
Keywords: TSC and LAM; Tuberous Sclerosis Complex and sporadic LAM
MeSH Terms: conditions — Tuberous Sclerosis; Lymphangioleiomyomatosis | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Rapamycin, sirolimus

SUMMARY:
The purpose of this study was to determine if rapamycin reduced angiomyolipomata volume in patients with tuberous sclerosis complex or lam.

DETAILED DESCRIPTION:
The study design was an open label, phase I/II trial of sirolimus for one year followed by one year off therapy.Patients were seen at baseline,at two weeks to four weeks, and at 2,4,6,9,12,18 and 24 months. Angiomyolipomata imaging was performed at all but the two to four week visit. Complete pulmonary function tests and six-minute walk were obtained at baseline,6 or 9 month, 12 and 24 month visits, while simple spirometry only was performed at all other visits.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with angiomyolipomas and have either Tuberous Sclerosis complex or Lymphangioleiomyomatosis
* Between the gaes of 18 and 65 years
* Competency to voluntarily consent
* Clinically definite diagnosis of tuberous sclerosis or S-LAM
* Adequate contraception
* At least one angiomyolipoma of 1 cm or greater in largest diameter

Exclusion Criteria:

* Use of continuous supplemental oxygen
* Concurrent infection
* Recent surgery
* Ongoing or planned pregnancy
* Lactation
* Use of an investigational drug within the last 30 days of study entrance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2002-12; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Volume of Angiomyolipomata

CONTACTS AND LOCATIONS:
Overall Officials: John Bissler, MD, Principal Investigator — Cincinnati Childrens Hospital Medical Center
Locations (1):
- Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Bissler JJ, McCormack FX, Young LR, Elwing JM, Chuck G, Leonard JM, Schmithorst VJ, Laor T, Brody AS, Bean J, Salisbury S, Franz DN. Sirolimus for angiomyolipoma in tuberous sclerosis complex or lymphangioleiomyomatosis. N Engl J Med. 2008 Jan 10;358(2):140-51. doi: 10.1056/NEJMoa063564. PMID 18184959